CLINICAL TRIAL: NCT01150747
Title: Chlamydia Trachomatis Immunology and Vaccinology Study: Determination of Protective T Cell Responses to Chlamydia Trachomatis Infection
Brief Title: Chlamydia Trachomatis Immunology and Vaccinology Study
Status: Completed | Type: Observational
Sponsor: Harold Wiesenfeld (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Harold Wiesenfeld, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO10010159; U19AI084024 (NIH)
Record Dates: First submitted 2010-06-23; First posted 2010-06-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Chlamydia
MeSH Terms: conditions — Chlamydia Infections | interventions — Ceftriaxone; Azithromycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Risk of positive chlamydia: 1. current, untreated endocervical C. trachomatis infection
  2. mucopurulent cervicitis on pelvic examination
  3. Sexual contact with a male partner recently diagnosed with C. trachomatis, and/or non-gonococcal urethritis
  Interventions: Drug: ceftriaxone; Drug: Azithromycin

INTERVENTIONS:
Drug: ceftriaxone — 250mg IM once
Drug: Azithromycin — 1 gm once

SUMMARY:
The primary objective is to prospectively follow 200 women with or at risk of cervicitis to determine the chlamydia-specific cellular responses that correlate with protection against incident infection. The hypothesis is that a positive IFN-y response by peripheral CD4+ T cells responding to stimulation with HSP60 will be significantly associated with protection from incident C. trachomatis infection.

DETAILED DESCRIPTION:
A total of 200 women with or at high risk of having cervicitis will be prospectively followed for correlations between chlamydia-specific cellular responses and protection against incident infection.

At enrollment participants will undergo a history and physical examination; blood draw; and pelvic examination including collection of vaginal and cervical samples, STD testing and endometrial biopsy.

Participants will have follow up visits conducted at 1, 4, 8 and 12 months following enrollment. At the follow-up visits, participants will undergo a repeat history and physical, blood draw and pelvic examination including collection of vaginal and cervical samples and STD testing.

The study design will allow comprehensive identification of the antigen-specific cell mediated immune responses most strongly associated with protection against C. trachomatis infection.

The primary objective is to prospectively follow 200 women with or at risk for cervicitis to determine the chlamydia-specific cellular responses that correlate with protection against incident infection.

ELIGIBILITY:
Inclusion Criteria

1. Women 15-35 years of age. Note: Minors must have written informed consent from her parent/legal guardian to participate.
2. At least one of the following:

   1. Current , untreated endocervical C. trachomatis infection.
   2. Mucopurulent cervicitis: defined by the presence of yellow or green endocervical mucopurulent discharge and/ or easily induced endocervical bleeding (bleeding when the first swab is placed in the endocervix).
   3. Sexual contact with a male partner (regardless of condom use) recently diagnosed (within the past 3 months) with C. trachomatis and/or non-gonococcal urethritis.

Exclusion Criteria:

1. Pregnant or nursing a baby. Note: a urine pregnancy test will be done at enrollment. Result must be negative to participate in the study.
2. Gynecologic surgery or surgical abortion in preceding 2 months of enrollment.
3. Allergy to any of the study medications and/or derivatives (cephalosporins, azithromycin, erythromycin, any macrolide or ketolide antibiotic) or Type 1 hypersensitivity allergic reaction to penicillin.
4. Systemic or vaginal antibiotic therapy in preceding 7 days of enrollment.
5. Prior hysterectomy.
6. Menopause.
7. Any condition, in the opinion of the investigator that would interfere with the participant's safety or with study outcomes.
8. Participation in any study involving an investigational product in the past 30 days or anticipation of participation in any study using an investigational product in the next 30 days.
9. Previous participation in this study.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women positive for chlamydia or at high risk of chlamydia infection.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Determination of the chlamydia-specific cellular responses that correlates with protection against incident infection | one year per patient

SECONDARY OUTCOMES:
Identify immunologic correlates associated with containment of the organism to the lower genital tract | one year per patient
Compare chlamydia-specific cellular responses in the PBMCs to endometrial lymphocytes | one year per patient
Evaluate the endocervical T cell phenotypes of women with containment of the organism to the lower genital tract | one year per patient
Characterize transcriptional inflammatory responses of women with Chlamydia | Study participation one year per patient
Use SNP analysis to identify genetic risk factors for chlamydia infection and disease | Study participation is one year per patient

CONTACTS AND LOCATIONS:
Overall Officials: Toni Darville, MD, Study Director — University of Pittsburgh
Locations (4):
- United States (4):
  - Allegheny County Sexually Transmitted Disease Clinic, Pittsburgh, Pennsylvania
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Mercy Hospital of UPMC, Pittsburgh, Pennsylvania